CLINICAL TRIAL: NCT05551117
Title: A Phase 2, Open-label, Study of Vobramitamab Duocarmazine in Participants With Metastatic Castration-resistant Prostate Cancer and Other Solid Tumors
Brief Title: A Study of Vobramitamab Duocarmazine in Participants With Metastatic Castration Resistant Prostate Cancer and Other Solid Tumors
Acronym: Tamarack
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGC018-03
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Castration-Resistant Prostatic Cancer; Androgen-Independent Prostatic Cancer; Androgen-Insensitive Prostatic Cancer; Androgen-Resistant Prostatic Cancer; Hormone Refractory Prostatic Cancer; Anal Cancer; Anal Neoplasm; Carcinoma, Squamous Cell of Head and Neck; Head and Neck Squamous Cell Carcinoma; Laryngeal Squamous Cell Carcinoma; Oral Squamous Cell Carcinoma; Malignant Melanoma; Melanoma; Non-small Cell Lung Cancer; Non-small Cell Carcinoma; Small-cell Lung Cancer; Small Cell Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Anus Neoplasms; Squamous Cell Carcinoma of Head and Neck; Melanoma; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Small Cell | interventions — abiraterone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: MGC018 2.0 mg (Arm A) (Experimental): MGC018 2.0 mg/kg every 4 weeks
  Interventions: Biological: vobramitamab duocarmazine 2.0 mg (Arm A)
- Part 1: MGC018 2.7 mg (Arm B) (Experimental): MGC018 2.7 mg/kg every 4 weeks
  Interventions: Biological: vobramitamab duocarmazine 2.7 mg (Arm B)
- Part 2 (Experimental): MGC018 2.7 mg/kg every 4 weeks
  Interventions: Biological: vobramitamab duocarmazine
- Part 1: Control Arm (Active Comparator): Patients are administered abiraterone or enzalutamide
  Interventions: Drug: Abiraterone; Drug: Enzalutamide

INTERVENTIONS:
Biological: vobramitamab duocarmazine 2.0 mg (Arm A) — 2.0 mg/kg intravenous (IV) every 4 weeks
  Other Names: MGC018
  Arms: Part 1: MGC018 2.0 mg (Arm A)
Biological: vobramitamab duocarmazine 2.7 mg (Arm B) — 2.7 mg.kg IV every 4 weeks
  Other Names: MGC018
  Arms: Part 1: MGC018 2.7 mg (Arm B)
Biological: vobramitamab duocarmazine — 2.7 mg.kg IV every 4 weeks
  Other Names: MGC018
  Arms: Part 2
Drug: Abiraterone — 1000 mg once daily
  Arms: Part 1: Control Arm
Drug: Enzalutamide — 160 mg daily
  Arms: Part 1: Control Arm

SUMMARY:
Study CP-MGC018-03 is an open-label, two-part, Phase 2 study. Part 1 of the study will enroll participants with metastatic castration-resistant prostate cancer (mCRPC) previously treated with one prior androgen receptor axis-targeted therapy (ARAT). ARAT includes abiraterone, enzalutamide, or apalutamide.

Participants may have received up to 1 prior docetaxel-containing regimen, but no other chemotherapy agents.

This part of the study will assess the efficacy and tolerability of vobramitamab duocarmazine (MGC018) in two experimental arms (2.0 mg/kg every 4 weeks [Q4W] and 2.7 mg/kg Q4W) . Approximately 100 participants will be randomized 1:1.

Part 2 of the study will enroll participants with locally advanced or metastatic solid tumors. Participants must have progressive following at least 1 prior line of standard chemotherapy for advanced or metastatic disease. Participants will receive vobramitamab duocarmazine at a dose of 2.7 mg/kg every 4 weeks. Up to 200 participants may be enrolled in Part 2.

In both parts, vobramitamab duocarmazine will be administered intravenously (IV) in clinic on Day 1 of each 4-week cycle. Vobramitamab duocarmazine will be administered until criteria for treatment discontinuation are met. Participants will undergo regular testing for signs of disease progression using computed tomography (CT) scans, magnetic resonance imaging (MRI), bone scans, and prostate-specific antigen (PSA) blood tests. Routine examinations and blood tests will be performed and evaluated by the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 only: Histologically confirmed adenocarcinoma of the prostate without evidence of neuroendocrine differentiation, signet cell, or small cell features.
* Part 2 only: Histologically confirmed SCC or the anus, melanoma, HNSCC, squamous NSCLC, or SCLC.
* Part 1 only: Received 1 prior ARAT for metastatic or non-metastatic, castration-sensitive or castration-resistant prostate cancer. A second ARAT regimen of <60 days used as bridging to lutetium-177 is permitted. Up to 3 total prior lines of therapy for mCRPC are permitted..
* Part 2 only: At least 1 prior line of systemic therapy for unresectable or metastatic disease and no more than 2 prior lines of cytotoxic chemotherapy. Participants with HNSCC or melanoma must have received prior PD-1 or PD-L1 inhibitor for advanced or metastatic disease.
* All participants must have ≥ 1 metastatic lesion, according to RECIST 1.1 or PCWG3 criteria, that is present on magnetic resonance imaging (MRI), computed tomography (CT), or bone scan obtained ≤ 28 days prior to initiation of study treatment.
* All participants must have tumor progression, according to disease-specific criteria, following their most recent anti-cancer therapy.
* All participants must have and available archival or formalin-fixed paraffin-embedded (FFPE) tumor tissue sample for participants with metastasis to internal organs
* All participants have acceptable physical condition and laboratory values.
* All participants of childbearing potential must agree to use highly effective methods of birth control.
* All participants must not be pregnant, planning to be pregnant, or breastfeeding.

Exclusion Criteria:

* Any underlying medical or psychiatric condition impairing participant's ability to receive, tolerate, or comply with the planned treatment or study procedures.
* Part 1 only: Received >1 prior taxane-containing regimen for prostate cancer. A second taxane regimen of <60 days used as bridging for lutetium-177 is permitted.
* Part 1 only: Received >3 total prior therapies for mCRPC
* Part 1 only: Participants with known BRCA or ATM mutation (germline or somatic) are not eligible unless they received prior treatment with a PARP inhibitor where available, indicated and tolerated.
* Another hematologic or solid tumor ≥ stage 1 malignancy that completed surgery, last dose of radiotherapy, or last dose of systemic anti-cancer therapy ≤ 2 years from first dose of study treatment. Participants who had curative therapy for non-melanomatous skin cancer or for localized malignancy are eligible.
* Untreated, symptomatic central nervous system (CNS) metastasis.
* Prior treatment with any B7-H3 targeted agent for cancer,
* Contradictions to the use of corticosteroid treatment
* Prior stem cell, tissue, or solid organ transplant.
* Part 1 only: Use of products that have published anti-prostate cancer activity or are known to decrease PSA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liudmila Schafer, M.D., Study Director — MacroGenics
Locations (63):
- United States (14):
  - Compassionate Cancer Care Medical Group, Fountain Valley, California
  - University of California Los Angeles (UCLA) Community Cancer Care, Los Angeles, California
  - The University of Florida Health System - UF Health Urology - Jacksonville, Jacksonville, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Pontchartrain Cancer Center, Covington, Louisiana
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute - Hudson-Webber Cancer Research Center, Detroit, Michigan
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Gabrail Cancer Center, Canton, Ohio
  - VA Portland Health Care Services, Portland, Oregon
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - Virginia Cancer Specalists, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (4):
  - Ramsay Health Care - Westmead Private Hospital, Westmead, New South Wales
  - The University of Queensland (UQ) - Princess Alexandra Hospital (PAH), Woolloongabba, Queensland
  - Cabrini Health- Malvern, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Belgium (5):
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Brussles
  - (Grand Hopital de Charleroi) GHDC, Charleroi, Hainaut
  - Centre Hospitalier de Ardenne - Libramont - Clinique du Sein, Libramont, Luxembourg
  - Centre Hospitalier Universitaire (CHU) - Universite Catholique de Louvain (UCL) - Namur - Site Godinne (Cliniques Universitaires UCL de Mont-Godinne), Godinne, Namur
  - Algemeen Ziekenhuis Maria Middelares, Ghent
- France (11):
  - Centre Antoine-Lacassagne, Nice, AM
  - Institut de Cancerologie Strasbourg Europe (ICANS), Strasbourg, Bas Rhin
  - Institut Bergonié, Bordeaux, Gironde
  - Institut régional du Cancer de Montpellier - ICM Val d'Aurelle, Montpellier, Herault
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire, Ille Et Vilaine
  - Clinique Victor Hugo, Le Mans, Sarthe
  - Gustave Roussy, Villejuif, Val De Marne
  - CHRU Brest, Brest
  - Institut Mutualiste Montsouris, Paris
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé, Île-de-France Region
  - Hopital Foch, Suresnes, Île-de-France Region
- Italy (5):
  - AOU San Luigi Gonzaga Oncology Department, Orbassano, TO
  - Ospedale dell'Angelo, Mestre, Venice
  - Radiation Oncology Unit, Azienda Ospedaliera Universitaria Careggi, University of Florence, Florence
  - Istituto Oncologico Veneto, Padua
  - Azienda Provinciale per i Servizi Sanitari - Presidio Ospedaliero S. Chiara, Trento
- Poland (6):
  - Szpital im. Fryderyka Chopina, Otwock, Masovian Voivodeship
  - Magodent Szpital Elblaska, Warsaw, Masovian Voivodeship
  - Medical Concierge Centrum Medyczne, Warsaw, Masovian Voivodeship
  - Grochowski Hospital, Warsaw, Masovian Voivodeship
  - Szpital Wojewodzki im. Mikolaja Kopernika, Koszalin, West Pomeranian Voivodeship
  - Przychodnia Lekarska "KOMED", Konin, WLKP
- South Korea (8):
  - Kyungpook National University Chilgok Hospital, Bugok, Daegu
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hopital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Samsung Meical Cemter, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (8):
  - Hospital Universitari Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville, Seville
  - Hospital Del Mar, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Institut Catala d'Oncologia Hospitalet, Barcelona
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - The Royal Marsden NHS Trust, Sutton, Surrey
  - Oxford University Hospitals NHS- Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: MGC018 2.0 mg (Arm A): vobramitamab duocarmazine 2.0 mg/kg, IV, every 4 weeks
- Part 1: MGC018 2.7 mg (Arm B): vobramitamab duocarmazine 2.7 mg/kg, IV, every 4 weeks
- Part 1: Control Arm: abiraterone 1000 mg once daily or enzalutamide 160 mg once daily.
- Part 2: vobramitamab duocarmazine 2.7 mg.kg, IV, every 4 weeks
Period: Overall Study
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Started | 91 | 90 | 7 | 4
Intent-to-treat Population | 91 | 90 | 7 | 4
Safety Population | 90 | 86 | 3 | 4
Tumor Response Evaluable Population | 59 | 49 | 3 | 4
Prostate-specific Antigen (PSA) Response Evaluable Population | 83 | 71 | 0 | 0
Anti-drug Antibody (ADA) Evaluable Population | 90 | 86 | 0 | 4
Completed | 58 | 56 | 2 | 2
Not Completed | 33 | 34 | 5 | 2
Not completed — Death | 23 | 20 | 0 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 13 | 4 | 0
Not completed — Elected to receive vobramitamab duocarmazine after protocol amendment 2. | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2 | Total
Number analyzed (Participants) | 91 | 90 | 7 | 4 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (9.03) | 69.1 (8.94) | 65.7 (10.47) | 51.8 (12.97) | 69.2 (9.45)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 3 | 3
  Male | 90 | 90 | 7 | 1 | 188
  Undifferentiated | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 0 | 0 | 19
  Not Hispanic or Latino | 47 | 50 | 6 | 4 | 107
  Unknown or Not Reported | 33 | 32 | 1 | 0 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 1 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 0 | 0 | 6
  White | 49 | 46 | 6 | 2 | 103
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 36 | 37 | 0 | 1 | 74
Region of Enrollment [Number; unit: participants]
  South Korea | 2 | 3 | 1 | 0 | 6
  Belgium | 4 | 5 | 0 | 0 | 9
  United States | 11 | 10 | 1 | 4 | 26
  Poland | 8 | 8 | 0 | 0 | 16
  Italy | 3 | 4 | 0 | 0 | 7
  United Kingdom | 6 | 4 | 4 | 0 | 14
  Australia | 4 | 1 | 1 | 0 | 6
  France | 35 | 35 | 0 | 0 | 70
  Spain | 18 | 20 | 0 | 0 | 38

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Six-month Radiographic Progression Free Survival (rPFS) as Determined by the Investigator
Description: The landmark analysis for 6 month rPFS rate will occur when all participants on Part 1 have been on study for at least 6 months.
Time Frame: Assessed every 8 weeks for six months. Six month data reported.
Population: All participants according to the study treatment assigned (Intent to Treat Population) for participants with mCRPC in Part 1 only. This outcome measure applies to Part 1 only. Per protocol, participants in Part 2 did not have mCRPC and were not part of this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Number analyzed (Participants) | 91 | 90 | 7 | 0
proportion of participants | 0.69 [0.57 to 0.78] | 0.70 [0.46 to 0.79] | 0.47 [0.021 to NA] — upper limit could not be estimated due to insufficient number of events. |

2. Primary Outcome: Part 2: Objective Response Rate (ORR) Per Investigator Assessment of Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 Criteria
Description: The ORR is defined as the percentage of participants in the response evaluable population who achieve a best overall response of complete response (CR) or partial response (PR), per RECIST version 1.1 criterial CR is defined as disappearance of all target and non-target lesions. PR is defined as at least a 30% decrease from baseline in the sum of diameters of target lesions.
Time Frame: Every 8 weeks for the first 24 weeks, then every 12 weeks. Average duration of participation, 10 months.
Population: All participants who received at least one dose of study treatment and had RECIST-evaluable disease per RECIST v1.1 (Tumor Response Evaluable Population) in Part 2 of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2
Number analyzed (Participants) | 4
percentage of participants | 0

3. Secondary Outcome: Part 1: ORR Per PCWG3 Criteria as Determined by the Investigator
Description: To qualify as an objective response, CR and PR require confirmation at least 4 weeks after initial observation of complete response (CR) or partial response (PR). CR + PR = ORR
Time Frame: Every 8 weeks for the first 24 weeks, then every 12 weeks. Average duration of participation, 10 months,
Population: The analysis is limited to only participants with mCRPC who experienced a complete or partial response to study treatment. None of the participants in the control arm experienced a complete or partial response to study treatment. Participants in Part 2 did not have mCRPC, so were not eligible for response using PCWG3 criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Number analyzed (Participants) | 59 | 49 | 3 | 0
percentage of participants | 13.6 | 30.6 | 0 |

4. Secondary Outcome: Part 1: Median Duration of Response (DoR) Per PCWG3 Criteria as Determined by the Investigator
Description: The DoR will be calculated as the time from the date of initial tumor response (CR or PR) to the date of first documented PD or death from any cause, whichever occurs first.
Time Frame: Every 8 weeks for the first 24 weeks, then every 12 weeks. Average duration of participation, 10 months.
Population: All participants with mCRPC who achieved a confirmed complete or partial response to study treatment. No participants in the control group had a complete or partial response. Participants in Part 2 did not have mCRPC, so were not eligible for response using PCWG3 criteria.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Number analyzed (Participants) | 8 | 15 | 0 | 0
months | 9.4 [3.68 to NA] — The upper bound of the CI could not be estimated due to insufficient number of participants with events | 9.1 [5.78 to 9.92] |  |

5. Secondary Outcome: Part 1: Mean Best Tumor Size Change Over Time
Time Frame: Every 8 weeks for the first 24 weeks, then every 12 weeks. Average duration of participation, 10 months.
Population: All participants with mCRPC who received at least one dose of study treatment and had RECIST-evaluable disease per PCWG3 (Tumor Response Evaluable Population) in Part 1 of the study. Participants in Part 2 of the study did not have mCRPC and are excluded from this analysis.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Number analyzed (Participants) | 59 | 49 | 2 | 0
percent change from baseline | -13.0 (59.70) | -29.0 (33.92) | -7.44 (7.16) |

6. Secondary Outcome: Part 1: Prostate-specific Cancer Antigen (PSA) Response Rate Per PCWG3 Criteria
Description: PSA response is defined as a ≥ 50% decline in PSA from baseline with PSA confirmation ≥ 3 weeks after the first documented reduction in PSA of ≥ 50%.
Time Frame: Every 4 weeks throughout study participation. Average duration 10 months.
Population: All participants in Part 1 who received at least one dose of study treatment, with a baseline PSA ≥ 2 ng/mL and at least one post-baseline PSA measurement (PSA Response Evaluable Population). There were no participants in the Control Arm that were part of the PSA Response Evaluable Population.
  Participants in Part 2 did not have mCRPC, so were not assessed using PSA measurement.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Number analyzed (Participants) | 83 | 71 | 0 | 0
percent | 45.8 [34.8 to 57.1] | 38.0 [26.8 to 50.3] |  |

7. Secondary Outcome: Part 1: Time to PSA Progression Per PCWG3 Criteria
Description: In participants with a decrease in PSA from baseline, PSA progression is defined as a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir value, which is confirmed by a consecutive second value obtained ≥ 3 weeks later.
  In participants with no decrease in PSA from baseline, PSA progression is defined as a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the baseline value after 12 weeks.
  Time to PSA progression is defined as the time from the date of randomization to the first PSA progression.
Time Frame: Every 4 weeks throughout study participation. Average duration of participation, 10 months.
Population: The ITT population for Part 1 was used for this analysis. Only 3 of 7 participants were treated in the in the control arm. Of the 3 participants treated in the control arm, only 1 participant had an event.
  Participants in Part 2 did not have mCRPC, so were not assessed using PSA measurement.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Number analyzed (Participants) | 91 | 90 | 1 | 0
months | 5.9 [4.63 to 6.97] | 6.9 [4.83 to NA] — The upper bound of the CI could not be estimated due to insufficient number of participants with event | 4.6 [NA to NA] — 95% confidence interval could not be calculated for 1 participant. |

8. Secondary Outcome: Part 1: Duration of PSA Response Per PCWG3 Criteria
Description: Duration of PSA response is defined as the time from the date of first documented PSA response to the earliest date of PSA progression.
Time Frame: Every 4 weeks throughout study participation. Average duration of participation, 10 months.
Population: All participants in Part 1 who met criteria for a PSA response to study treatment. There were no participants in the Control Arm that were part of the PSA Response Evaluable Population. Participants in Part 2 did not have mCRPC, so were not assessed using PSA measurement.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Number analyzed (Participants) | 38 | 27 | 0 | 0
months | 6.1 [4.63 to NA] — The upper bound of the CI could not be estimated due to insufficient number of participants with event | NA [5.13 to NA] — The median and upper bound of the CI could not be estimated due to insufficient number of participants with events |  |

9. Secondary Outcome: Part 1: Best PSA Percent Change
Time Frame: Every 4 weeks throughout study participation. Average duration of participation, 10 months.
Population: PSA Response Evaluable Population. There were no participants in the Control Arm that were part of the PSA Response Evaluable Population. Participants in Part 2 did not have mCRPC, so were not assessed using PSA measurement.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Number analyzed (Participants) | 83 | 71 | 0 | 0
percent change from baseline | -28.7 (67.05) | -33.1 (70.89) |  |

10. Secondary Outcome: Part 1: Time to First Symptomatic Skeletal Event (SSE)
Description: An SSE is defined as any of the following events: new symptomatic pathological fracture, requirement for radiation therapy to relieve bone pain, spinal cord compression, or tumor-related orthopedic surgical intervention. The time to first SSE is defined as the time from the date of randomization to the first occurrence of SSE.
Time Frame: Every 4 weeks throughout the study. Average duration of participation, 10 months.
Population: Participants who experienced a symptomatic skeletal event in Part 1 of the study. SSE were not assessed in Part 2, as these participants did not have mCRPC.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Number analyzed (Participants) | 5 | 7 | 0 | 0
days | 3.71 (1.984) | 2.80 (2.142) |  |

11. Secondary Outcome: Number of Participants With Adverse Event (AEs), Serious AEs (SAEs), and AEs Leading to Study Treatment Discontinuation.
Time Frame: Throughout the study, average duration of participation, 10 months.
Population: The Safety Population was used for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Number analyzed (Participants) | 90 | 86 | 3 | 4
Participants
  Any Adverse Event | 89 | 86 | 3 | 4
  Serious Adverse Events | 36 | 44 | 1 | 2
  Adverse Events Leading to Discontinuation | 28 | 41 | 0 | 2

12. Secondary Outcome: Number of Participants Who Develop Anti-drug Antibodies (ADA)
Description: Participant specimens were evaluated for the presence of ADA beginning a baseline and throughout the study. If at any time during the study, the results show evidence of ADA, they were counted as ADA positive. There was no time-to- event analysis nor by visit analysis of the data.
Time Frame: Every 4 weeks throughout the study, average duration of participation was 10 months.
Population: The ADA Evaluable Population was used for this analysis. Participants in the control arm did not receive MGC018.
Measure: Number; unit: participants
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
Number analyzed (Participants) | 90 | 86 | 0 | 4
participants
  Positive ADA at baseline | 0 | 0 |  | 0
  Positive ADA at any time after dosing. | 22 | 16 |  | 0

13. Secondary Outcome: Part 2: Median DoR Per Investigator Assessment of RECIST 1.1 Criteria
Description: The DoR will be calculated as the time from the date of initial tumor response (CR or PR) to the date of first documented progressive disease (PD) or death from any cause, whichever occurs first.
Time Frame: Every 8 weeks for the first 24 weeks, then every 12 weeks. Average duration of participation, 10 months.
Population: No participants in Part 2 of the study had a complete or partial response to study treatment.
Arm/Group | Part 2
Number analyzed (Participants) | 0

14. Secondary Outcome: Part 2: Median Progression Free Survival (PFS) Per Investigator Assessment of RECIST 1.1 Criteria
Description: PFS is defined as the time from the date of the first dose to the date of first PD per RECIST 1.1 criteria or death from any cause, whichever occurs first.
Time Frame: Every 8 weeks for the first 24 weeks, then every 12 weeks. Average duration of participation, 10 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2
Number analyzed (Participants) | 4
months | NA [NA to NA] — Cannot be estimated due to insufficient number of events.

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from the time of first dose through 28 days after the last dose of study treatment or until the start of another anti-cancer treatment, up to average duration of participation, 10 months months. All-cause mortality was assessed from the time of first dose until death, or participant withdrawal of consent, or the end of the study, whichever was earlier, up to average duration of participation, 10 months.
Description: Adverse events are based on physical findings, patient reports, and significant laboratory values.
  Progression of neoplasm causing hospitalization or death is an antitumor activity outcome and not an SAE, unless considered drug-related by the investigator.
Arm/Group | Part 1: MGC018 2.0 mg (Arm A) | Part 1: MGC018 2.7 mg (Arm B) | Part 1: Control Arm | Part 2
All-Cause Mortality (participants affected / at risk) | 25/90 | 21/86 | 1/3 | 2/4
Serious Adverse Events (participants affected / at risk) | 36/90 | 44/86 | 1/3 | 2/4
Other Adverse Events (participants affected / at risk) | 89/90 | 86/86 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: MGC018 2.0 mg (Arm A) (N=90) | Part 1: MGC018 2.7 mg (Arm B) (N=86) | Part 1: Control Arm (N=3) | Part 2 (N=4)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 5 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 4 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Hypothalamo-pituitary disorder (Endocrine disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Overflow diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 2 | 3 | 0 | 0
Generalised oedema (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 5 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Oral infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Thrombophlebitis septic (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Calcium deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 12 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: MGC018 2.0 mg (Arm A) (N=90) | Part 1: MGC018 2.7 mg (Arm B) (N=86) | Part 1: Control Arm (N=3) | Part 2 (N=4)
Anaemia (Blood and lymphatic system disorders) | 19 | 23 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 17 | 22 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 12 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 4 | 10 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 8 | 0 | 0
Pericardial effusion (Cardiac disorders) | 13 | 13 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 4 | 0 | 0
Dry eye (Eye disorders) | 10 | 10 | 0 | 1
Eyelid oedema (Eye disorders) | 6 | 9 | 0 | 0
Lacrimation increased (Eye disorders) | 5 | 5 | 0 | 0
Nausea (Gastrointestinal disorders) | 32 | 26 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 26 | 20 | 0 | 0
Constipation (Gastrointestinal disorders) | 22 | 20 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 13 | 23 | 0 | 0
Vomiting (Gastrointestinal disorders) | 15 | 5 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 9 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 8 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 7 | 3 | 0 | 1
Asthenia (General disorders) | 47 | 52 | 0 | 0
Oedema peripheral (General disorders) | 33 | 35 | 0 | 1
Fatigue (General disorders) | 25 | 20 | 2 | 2
Pyrexia (General disorders) | 11 | 12 | 0 | 0
Chills (General disorders) | 5 | 7 | 0 | 0
Face oedema (General disorders) | 7 | 2 | 0 | 1
Conjunctivitis (Infections and infestations) | 11 | 17 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 5 | 0 | 0
Herpes zoster (Infections and infestations) | 4 | 6 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 11 | 0 | 0
Weight decreased (Investigations) | 10 | 9 | 0 | 1
Platelet count decreased (Investigations) | 7 | 8 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 5 | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 6 | 0 | 1
White blood cell count decreased (Investigations) | 5 | 4 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 33 | 35 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 6 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 7 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 10 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 8 | 0 | 0
Headache (Nervous system disorders) | 12 | 16 | 0 | 2
Dysgeusia (Nervous system disorders) | 10 | 11 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 9 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 10 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 25 | 29 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 16 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 13 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 | 24 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 11 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 7 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 | 5 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT05551117/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT05551117/SAP_001.pdf